CLINICAL TRIAL: NCT05509114
Title: The Effect of Virtual Reality Glasses Application on Pain, Anxiety, and Patient Satisfaction During a Transrectal Prostate Biopsy: A Randomized Controlled Trial
Brief Title: The Effect of Virtual Reality Glasses Application on Pain, Anxiety, and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Rumeysa Lale TORAMAN, Research Assistant, Ataturk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Rumeysa
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Prostate
Keywords: anxiety, pain, patient satisfaction, virtual reality
MeSH Terms: conditions — Anxiety Disorders; Pain; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Glasses (Experimental): The intervention introductory information formula was face-to-face by researchers from the State-Trait Anxiety Inventory (STAI-I, STAI-II), the Scale of Patient Perception of Hospital Experience with Nursing Care (PPHEN) and Visual Analog Scale for Pain (VAS) Before starting the research, a preliminary application plan is determined with 10 virtual virtual applications. It is not included in the applications made in the pre-application. Before watching the video, patients are informed about how to train, how to do it, and detailed information about the video. When the patient is removed from the service and in the left lateral position, 2 minutes before the assistant physician, the virtual is about to take place. The video was watched after about 10-15 minutes until the process was finished. After the procedure, STAI-I, STAI-II, PPHEN and VAS were reapplied by the researchers.
  Interventions: Device: Virtual Reality Glasses

INTERVENTIONS:
Device: Virtual Reality Glasses — The intervention group of patients watched a video with virtual reality glasses during the transrectal biopsy process.

SUMMARY:
The study was conducted in a randomized controlled manner to determine the effect of applying virtual reality glasses during transrectal prostate biopsy on pain, anxiety and patient satisfaction.The study was completed with a total of 70 patients, 35 in the intervention group and 35 in the control group, for whom it was decided to perform sample transrectal prostate biopsy for the first time.

DETAILED DESCRIPTION:
Although prostate cancer is the most common type of cancer in men, according to 2018 data published by the International Agency for Research on Cancer, it is the second most common after lung cancer worldwide.The prevalence of prostate cancer is increasing rapidly worldwide. However, when prostate cancer is diagnosed early, the survival rate increases with the effect of the treatment methods applied. Digital rectal examination (DRE), prostate specific antigen (PSA) level, and transrectal ultrasonography-guided prostate biopsy (TRUS-Bx) methods are used for diagnosis. Transrectal prostate biopsy process; It is one of the most frequently performed urological procedures for definitive diagnosis in patients with a PSA value above the normal limit and abnormal DRE findings. Transrectal prostate biopsy is a golden diagnostic tool in prostate cancer because it is typically well tolerated, treatable, and has a low risk of major complications. However, in addition to the advantages of this procedure, it also has disadvantages such as causing pain and discomfort in patients.Prostate biopsy procedure affects patients not only physiologically but also psychologically. Interventional procedures cause patients to experience the highest level of anxiety. With the development of technology, developments in health care have brought the concept of patient satisfaction to the fore. Applications made in line with patient expectations in order to increase the quality of care make a significant contribution to the perception of nursing care. One of these applications, virtual reality glasses, make patients feel like they are in a different world; increases patient satisfaction. Nurses, who are members of the profession who plan and manage care, because they spend longer time with the patient; They play an active role in defining pain and anxiety by using pharmacological and non-pharmacological methods. When examining the literature, there was no study examining the effect of virtual reality application on the pain level of patients during the transrectal prostate biopsy procedure, but no study examining the effect on the level of anxiety and patient satisfaction. In this study; It is aimed to increase patient satisfaction by reducing the pain and anxiety of the patients with virtual reality applied during the transrectal prostate biopsy procedure. It is thought that the results of this study can make an important contribution to both the literature and practice.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18-65,
* Those who volunteer and accept to participate in the research,
* Transrectal prostate biopsy procedure performed for the first time,
* No communication problem,
* Cognitive level scales are suitable for application,
* Patients without vision or hearing problems were included in the study.

Exclusion Criteria:

* Leaving work voluntarily,
* Patients whose cognitive level scales were not suitable for application were excluded from the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-12-25 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety İnventory (STAI-I, STAI-II) | up to 24 hours
  It is a test developed by Spielberger et al. that measures state and trait anxiety levels. Its validity and reliability in Turkey was done by Öner and Le Compte. The scale consists of two parts, the 'state anxiety scale', which is created with the aim of determining the instantaneous feelings, and the 20-item 'trait anxiety scale', which was created to determine the feelings in general. It is a four degree scale ranging from 'Nothing' to 'All'. Scores range from 20 (low anxiety) to 80 (high anxiety).
The Scale of Patient Perception of Hospital Experience with Nursing Care (PPHEN) | up to 24 hours
  The patient's perception of nursing care scale was developed by Dozier et al. in the USA, and its Turkish validity and reliability were determined by Çoban and Kaşıkçı.Likert-type scale has 15 statements about the quality of nursing care. A minimum of 15 and a maximum of 75 points can be obtained from the scale. The cut-off point of the scale is 45. Scores above the cut-off point indicate a positive attitude. The increase in the total score obtained from the scale indicates that the patient is satisfied with the nursing care.
Visual Analog Scale for Pain (VAS) | up to 24 hours
  VAS is a scale developed by Price et al34 (1983) and measures the severity of pain in the patient. VAS is a 10 cm long vertical or horizontal scale with two different names (0=no pain, 10=most severe pain). An increase in the score obtained from the scale in the evaluation indicates an increase in pain.

CONTACTS AND LOCATIONS:
Overall Officials: Rumeysa Lale TORAMAN, Principal Investigator — Ataturk University
Locations (1):
- Rumeysa Lale TORAMAN, Palandöken, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No